CLINICAL TRIAL: NCT03138889
Title: A Phase 1/2, Open-Label, Multicenter Study to Investigate the Safety and Preliminary Efficacy of Combined Bempegaldesleukin (NKTR-214) and Pembrolizumab With or Without Chemotherapy in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Bempegaldesleukin and Pembrolizumab With or Without Chemotherapy in Locally Advanced or Metastatic Solid Tumors
Acronym: PROPEL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-214-05
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NKTR-214; Metastatic Non-Small Cell Lung Cancer; Pembrolizumab; Keytruda®; NSCLC; Bempegaldesleukin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — bempegaldesleukin; pembrolizumab; Cisplatin; Carboplatin; Taxes; Albumin-Bound Paclitaxel; Paclitaxel; Pemetrexed; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Optimization, Combo of NKTR-214 + Pembrolizumab(KEYTRUDA®) (Experimental): Cohort 1: NKTR-214 will be combined with pembrolizumab
  Interventions: Drug: NKTR-214; Drug: Pembrolizumab
- Dose Expansion, Combo of NKTR-214 + Pembrolizumab(KEYTRUDA®) (Experimental): Cohort 2: NKTR-214 will be combined with pembrolizumab
  Interventions: Drug: Pembrolizumab; Drug: NKTR-214
- Dose Expansion, Combo of NKTR-214 + Pembrolizumab (KEYTRUDA®) (Experimental): Cohort 3: NKTR-214 will be combined with pembrolizumab
  Interventions: Drug: Pembrolizumab; Drug: NKTR-214
- Dose Expansion, NKTR-214 + Pembrolizumab and either Cisplatin, or Carboplatin and Pemetrexed (Experimental): Cohort 4: NKTR-214 will be dosed in combination with pembrolizumab and either cisplatin, or carboplatin and pemetrexed, per investigator discretion
  Interventions: Drug: Pembrolizumab; Drug: NKTR-214; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed
- Dose Expansion, NKTR-214 + Pembrolizumab and Carboplatin and either Nab-paclitaxel or Paclitaxel (Experimental): Cohort 5: NKTR-214 will be dosed in combination with pembrolizumab and carboplatin and either nab-paclitaxel or paclitaxel, per investigator discretion
  Interventions: Drug: Pembrolizumab; Drug: NKTR-214; Drug: Carboplatin; Drug: Nab paclitaxel; Drug: Paclitaxel
- Combo of NKTR-214 + Pembrolizumab(KEYTRUDA®) or Atezolizumab (TECENTRIQ®) (Experimental): Cohort 0 (Before Protocol Amendment 5.0): NKTR-214 will be combined with pembrolizumab or atezolizumab
  Interventions: Drug: Pembrolizumab; Drug: NKTR-214; Drug: Atezolizumab

INTERVENTIONS:
Drug: NKTR-214 — NKTR-214: The dose will be 0.008 mg/kg intravenous (IV) infusion administered over 30 (± 5) minutes q3w. The maximum dose of NKTR-214 will be 0.012 mg/kg. This will include a fixed 3+3 dose escalation followed by intra-patient step-up dose escalation based on tolerability.
  Other Names: CD122-Biased Cytokine
  Arms: Dose Optimization, Combo of NKTR-214 + Pembrolizumab(KEYTRUDA®)
Drug: Pembrolizumab — Pembrolizumab (anti-PD-1) will be dosed as per the pharmacy manual.
  Other Names: Keytruda®
Drug: NKTR-214 — NKTR-214: The dose will be 0.006 mg/kg intravenous (IV) infusion.
  Other Names: CD122-Biased Cytokine
  Arms: Combo of NKTR-214 + Pembrolizumab(KEYTRUDA®) or Atezolizumab (TECENTRIQ®); Dose Expansion, Combo of NKTR-214 + Pembrolizumab(KEYTRUDA®); Dose Expansion, NKTR-214 + Pembrolizumab and Carboplatin and either Nab-paclitaxel or Paclitaxel; Dose Expansion, NKTR-214 + Pembrolizumab and either Cisplatin, or Carboplatin and Pemetrexed
Drug: NKTR-214 — NKTR-214: The dose will be 0.010 mg/kg intravenous (IV) infusion.
  Other Names: CD122-Biased Cytokine
  Arms: Dose Expansion, Combo of NKTR-214 + Pembrolizumab (KEYTRUDA®)
Drug: Cisplatin — Cisplatin will be dosed per the pharmacy manual
  Other Names: Platinol®
  Arms: Dose Expansion, NKTR-214 + Pembrolizumab and either Cisplatin, or Carboplatin and Pemetrexed
Drug: Carboplatin — Carboplatin will be dosed per the pharmacy manual
  Other Names: Paraplatin®
  Arms: Dose Expansion, NKTR-214 + Pembrolizumab and Carboplatin and either Nab-paclitaxel or Paclitaxel; Dose Expansion, NKTR-214 + Pembrolizumab and either Cisplatin, or Carboplatin and Pemetrexed
Drug: Nab paclitaxel — Nab-paclitaxel will be dosed per local practice and label
  Other Names: Abraxane®
  Arms: Dose Expansion, NKTR-214 + Pembrolizumab and Carboplatin and either Nab-paclitaxel or Paclitaxel
Drug: Paclitaxel — Paclitaxel will be dosed per local practice and label
  Other Names: Taxol®
  Arms: Dose Expansion, NKTR-214 + Pembrolizumab and Carboplatin and either Nab-paclitaxel or Paclitaxel
Drug: Pemetrexed — Pemetrexed will be dosed per the pharmacy manual
  Other Names: Alimta®
  Arms: Dose Expansion, NKTR-214 + Pembrolizumab and either Cisplatin, or Carboplatin and Pemetrexed
Drug: Atezolizumab — Atezolizumab will be dosed per current label indication
  Other Names: Tecentriq®
  Arms: Combo of NKTR-214 + Pembrolizumab(KEYTRUDA®) or Atezolizumab (TECENTRIQ®)

SUMMARY:
This study is to assess the safety and tolerability, and to assess the preliminary clinical benefit of NKTR-214 when combined with pembrolizumab (KEYTRUDA®) with or without chemotherapy.

The study is comprised of two groups; dose optimization and dose expansion cohorts.

Dose Optimization included first-line and second-line advanced or metastatic solid tumors including non-small cell lung cancer (NSCLC)

The dose expansion cohort will include first-line NSCLC patients.

DETAILED DESCRIPTION:
NKTR-214 is a cytokine (investigational agent) that is designed to target CD122, a protein which is found on certain immune cells (known as CD8+ T Cells and Natural Killer Cells) to expand these cells to promote their anti-tumor effects. Pembrolizumab is a programmed death receptor -1 (PD-1) blocking, fully humanized, engineered monoclonal antibody of IgG1 isotype that promotes anti-tumor effects.

The study will evaluate the clinical benefit, safety and tolerability of combining NKTR-214 with pembrolizumab with or without chemotherapy. Each dose expansion cohort will enroll approximately 100 new patients.

Dose Optimization evaluated an every three-week dose regimen (q3w) of NKTR-214 in combination with pembrolizumab given that the optimal dose and dosing schedule of NKTR-214 in combination with pembrolizumab remains unknown. The previously established recommended Phase 2 dose (0.006 mg/kg) of NKTR-214 was studied in combination with nivolumab.

Dose Expansion: NKTR-214 in combination with pembrolizumab will be evaluated in first-line non-small cell lung cancer (NSCLC). The NKTR-214 dose to be studied is 0.006 mg/kg q3w. This dose is based on the recommended phase 2 dose noted in the monotherapy trial with NKTR-214 (Study 15-214-01, NCT02869295) and an ongoing combination trial (16-214-02, NCT02983045). Pembrolizumab will be administered at a dose of 200mg q3w. Following data review for safety and efficacy, additional patients may be dosed using the findings from the dose optimization cohorts.

ELIGIBILITY:
Inclusion Criteria:

Dose Optimization and Dose Expansion Inclusion Criteria:

* Willing and able to provide written informed consent.
* Male or female patients, age 18 years or older at the time of signing the informed consent form (ICF).
* Life expectancy > 12 weeks from the time of enrollment as determined by the Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Oxygen saturation ≥ 92% on room air for all indications.
* Measurable disease per RECIST 1.1.
* Patients with brain metastases are eligible if certain criteria are met.
* Availability of fresh or archival tumor tissue
* Patients must have a minimum of 6 months of response to any nonpalliative cancer-directed treatment

Dose Expansion Inclusion Criteria (Non-Small Cell Lung Cancer):

* Histologically confirmed diagnosis of stage IV NSCLC.
* Patients must have a minimum of 6 months of response to any nonpalliative cancer-directed treatment.
* Patients with actionable mutations with approved targeted therapy in NSCLC are excluded. Testing for mutations should be performed per standard of care.
* Must not have received anti-cancer therapy for treatment of metastatic lung cancer
* Must not have received prior immunotherapy

Exclusion Criteria:

* Use of an investigational agent or an investigational device within 28 days before administration of first dose of study drug(s).
* Females who are pregnant or breastfeeding.
* Patients who have an active autoimmune disease
* History of allergy or hypersensitivity to study drug components
* Evidence of clinically significant interstitial lung disease or active, noninfectious pneumonitis.
* Prior surgery or radiotherapy within 14 days of therapy.
* For Dose Optimization Cohort 1 only: Chemotherapy or biological therapy within 28 days of enrollment. Targeted therapy (e.g., tyrosine kinase inhibitors) within 14 days of enrollment. Patients with ongoing AEs related to prior cancer therapies will be excluded.
* Participant's inability to adhere to or tolerate protocol or study procedures

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (38):
- United States (23):
  - Highlands Oncology Group, PA - North Hills, Fayetteville, Arkansas
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Augusta University - Augusta University Medical Center, Augusta, Georgia
  - Ochsner Medical Center, New Orleans, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Park Nicollet - Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada (CCCN) - Central Valley, Las Vegas, Nevada
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke Clinical Research Institute, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - West Cancer Center, Germantown, Tennessee
  - Sarah Cannon Research Institute (SCRI) (The SCRI Oncology Research Consortium), Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Inova Melanoma and Skin Cancer Center, Fairfax, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
  - Froedtert & the Medical College of Wisconsin Froedtert Hospital, Milwaukee, Wisconsin
- Epworth HealthCare, Richmond, Victoria, Australia
- Centre Hospitalier de Saint-Quentin, Saint-Quentin, France
- Germany (6):
  - Vivantes Klinikum Spandau, Berlin
  - Asklepios Fachkliniken München-Gauting, Gauting
  - LungenClinic Grosshansdorf, Großhansdorf
  - Lungenklinik Hemer, Hemer
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Robert-Bosch-Krankenhaus, Stuttgart
- Spain (7):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - HM Universitario Sanchinarro, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 0 (Before Protocol Amendment 5.0): NKTR-214 (0.006 mg/kg) + Pembro (200 mg): NKTR-214 (0.006 mg/kg) every 3 weeks (q3w) + pembrolizumab 200 mg
  NKTR-214: Specified dose on specified days Pembrolizumab: Specified dose on specified days
- Cohort 0 (Before Protocol Amendment 5.0): NKTR-214 (0.006 mg/kg) + Atezo (1200 mg): NKTR-214 (0.006 mg/kg) every 3 weeks (q3w) + atezolizumab 1200 mg
  NKTR-214: Specified dose on specified days Atezolizumab: Specified dose on specified days
- Dose Optimization Cohort 1a: NKTR-214 (0.008 mg/kg) + Pembro (200 mg): NKTR-214 (0.008 mg/kg) q3w + pembrolizumab (200 mg)
  NKTR-214: Specified dose on specified days Pembrolizumab: Specified dose on specified days
- Dose Optimization Cohort 1a: NKTR-214 (0.010 mg/kg) + Pembro (200 mg): NKTR-214 (0.010 mg/kg) q3w + pembrolizumab (200 mg)
  NKTR-214: Specified dose on specified days Pembrolizumab: Specified dose on specified days
- Dose Optimization Cohort 1a: NKTR-214 (0.012 mg/kg) + Pembro (200 mg): NKTR-214 (0.012 mg/kg) q3w + pembrolizumab (200 mg)
  NKTR-214: Specified dose on specified days Pembrolizumab: Specified dose on specified days
- Dose Expansion Cohort 2: NKTR-214 (0.006 mg/kg) + Pembro (200 mg): NKTR-214 (0.006 mg/kg) + pembrolizumab (200 mg)
  NKTR-214: Specified dose on specified days Pembrolizumab: Specified dose on specified days
- Dose Expansion Cohort 3: NKTR-214 (0.010 mg/kg) + Pembro (200 mg): NKTR-214 (0.010 mg/kg) + pembrolizumab (200 mg)
  NKTR-214: Specified dose on specified days Pembrolizumab: Specified dose on specified days
- Dose Expansion Cohorts 4/5: NKTR-214 (0.006 mg/kg) + Pembro (200 mg) + Chemotherapy: NKTR-214 (0.006 mg/kg) + pembrolizumab (200 mg) + chemotherapy
  NKTR-214: Specified dose on specified days Pembrolizumab: Specified dose on specified days
Period: Overall Study
Arm/Group | Cohort 0 (Before Protocol Amendment 5.0): NKTR-214 (0.006 mg/kg) + Pembro (200 mg) | Cohort 0 (Before Protocol Amendment 5.0): NKTR-214 (0.006 mg/kg) + Atezo (1200 mg) | Dose Optimization Cohort 1a: NKTR-214 (0.008 mg/kg) + Pembro (200 mg) | Dose Optimization Cohort 1a: NKTR-214 (0.010 mg/kg) + Pembro (200 mg) | Dose Optimization Cohort 1a: NKTR-214 (0.012 mg/kg) + Pembro (200 mg) | Dose Expansion Cohort 2: NKTR-214 (0.006 mg/kg) + Pembro (200 mg) | Dose Expansion Cohort 3: NKTR-214 (0.010 mg/kg) + Pembro (200 mg) | Dose Expansion Cohorts 4/5: NKTR-214 (0.006 mg/kg) + Pembro (200 mg) + Chemotherapy
Started | 12 | 23 | 4 | 7 | 7 | 75 | 17 | 17
Completed | 7 | 18 | 4 | 5 | 6 | 72 | 17 | 16
Not Completed | 5 | 5 | 0 | 2 | 1 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 5 | 0 | 2 | 1 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: * Safety population: all patients who received at least one dose (or partial dose) of study treatment
  * Dose-limiting toxicity (DLT) Population: all patients who completed at least the DLT observation period or discontinued from the study treatment due to DLT
  * Response evaluable population: subjects who received at least 1 dose (or partial dose) of study drug, had measurable disease (per RECIST 1.1) at baseline, and had at least one post-baseline assessment of tumor response.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 0 (Before Protocol Amendment 5.0): NKTR-214 (0.006 mg/kg) + Pembro (200 mg) | Cohort 0 (Before Protocol Amendment 5.0): NKTR-214 (0.006 mg/kg) + Atezo (1200 mg) | Dose Optimization Cohort 1a: NKTR-214 (0.008 mg/kg) + Pembro (200 mg) | Dose Optimization Cohort 1a: NKTR-214 (0.010 mg/kg) + Pembro (200 mg) | Dose Optimization Cohort 1a: NKTR-214 (0.012 mg/kg) + Pembro (200 mg) | Dose Expansion Cohort 2: NKTR-214 (0.006 mg/kg) + Pembro (200 mg) | Dose Expansion Cohort 3: NKTR-214 (0.010 mg/kg) + Pembro (200 mg) | Dose Expansion Cohorts 4/5: NKTR-214 (0.006 mg/kg) + Pembro (200 mg) + Chemotherapy | Total
Number analyzed (Participants) | 12 | 23 | 4 | 7 | 7 | 75 | 17 | 17 | 162
Age, Customized [Number; unit: participants]
  Age < 65 | 5 | 11 | 2 | 3 | 3 | 35 | 6 | 9 | 74
  Age 65-84 | 6 | 12 | 2 | 4 | 4 | 40 | 11 | 8 | 87
  Age 85 and Over | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 2 | 4 | 5 | 24 | 4 | 7 | 57
  Male | 7 | 17 | 2 | 3 | 2 | 51 | 13 | 10 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 5
  Not Hispanic or Latino | 11 | 19 | 4 | 7 | 7 | 65 | 17 | 14 | 144
  Unknown or Not Reported | 1 | 2 | 0 | 0 | 0 | 7 | 0 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 7
  White | 10 | 21 | 4 | 7 | 6 | 72 | 16 | 15 | 151
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 12 | 23 | 4 | 7 | 7 | 25 | 3 | 15 | 96
  Italy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  France | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Germany | 0 | 0 | 0 | 0 | 0 | 16 | 2 | 2 | 20
  Spain | 0 | 0 | 0 | 0 | 0 | 32 | 12 | 0 | 44
ECOG [Count of Participants; unit: Participants] — Measure Description: Eastern Cooperative Oncology Group (ECOG) performance status:
  ECOG Performance Status of 0 = Able to carry out all normal activities without restriction ECOG Performance Status of 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature
  Participants
    ECOG 0 | 7 | 11 | 3 | 2 | 5 | 33 | 8 | 6 | 75
    ECOG 1 | 5 | 12 | 1 | 5 | 2 | 42 | 9 | 11 | 87

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-Limiting Toxicities in Dose Optimization Cohort 1a
Description: DLTs were assesses in the Dose Optimization Cohort 1 a, which had doses of NKTR-214 as 0.008 mg/kg, 0.010 mg/kg, and 0.012 m/kg, I combination with pembrolizumab at 200 mg.
  A single DLT (hypotension) was reported in 1 patient in dose optimization Cohort 1a.
Time Frame: DLTs were assessed at 21 days from Cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Optimization Cohort 1a: NKTR-214 (0.008 mg/kg) + Pembro (200 mg) | Dose Optimization Cohort 1a: NKTR-214 (0.010 mg/kg) + Pembro (200 mg) | Dose Optimization Cohort 1a: NKTR-214 (0.012 mg/kg) + Pembro (200 mg)
Number analyzed (Participants) | 4 | 7 | 7
Participants
  At least 1 DLT | 0 | 1 | 0
  Vascular Disorders: Hypotension | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events [Safety and Tolerability] for Dose Optimization Cohort 1a.
Description: Safety and Tolerability of NKTR-214 (starting at dose of 0.008 mg/kg) in combination with pembrolizumab (Keytruda®) as evaluated by incidence of drug-emergent Adverse Events (AEs), Serious Adverse Events (SAEs), AEs leading to drug discontinuation, and fatal AEs.
Time Frame: AEs reported starting immediately after first dose of study drug(s) until 100 days after the last dose of all study drugs, up to approximately 28 months.
Measure: Count of Participants; unit: Participants
Groups:
- NKTR-214 (0.008 mg/kg) + Pembro (200 mg): NKTR-214 0.008 mg/kg every 3 weeks + pembrolizumab 200 mg
- NKTR-214 (0.010 mg/kg) + Pembro (200 mg): NKTR-214 0.010 mg/kg every 3 weeks + pembrolizumab 200 mg
- NKTR-214 (0.012 mg/kg) + Pembro (200 mg): NKTR-214 0.012 mg/kg every three weeks + pembrolizumab 200 mg
- Total: Total (N=18)
Arm/Group | NKTR-214 (0.008 mg/kg) + Pembro (200 mg) | NKTR-214 (0.010 mg/kg) + Pembro (200 mg) | NKTR-214 (0.012 mg/kg) + Pembro (200 mg) | Total
Number analyzed (Participants) | 4 | 7 | 7 | 18
Participants
  Subjects Reporting at Least One TEAE | 4 | 7 | 7 | 18
  Subjects Reporting at Least One Serious TEAE | 2 | 4 | 2 | 8
  Subjects Reporting at Least One TEAE Leading to Death | 0 | 0 | 0 | 0
  Subjects Reporting at Least One TEAE Leading to Drug Discontinuation | 2 | 3 | 1 | 6

3. Primary Outcome: Objective Response Rate (ORR) Per Blinded Independent Central Review (BICR) by RECIST 1.1 of NKTR-214 Plus Pembrolizumab for Dose Expansion Cohorts 2 and 3.
Description: ORR per BICR by RECIST 1.1 for the Response Evaluable Population dose expansion Cohorts 2 and 3.
  ORR is defined as the proportion of enrolled participants who achieved a Best Overall Response (BOR) of CR or PR. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR is calculated as the sum of CR and PR.
  The Response Evaluable Population was subjects who received at least 1 dose (or partial dose) of study drug, had measurable disease (per RECIST 1.1) at baseline, and had at least 1 post-baseline assessment of tumor response.
Time Frame: Until disease progression, death, unacceptable toxicity, symptomatic deterioration, Investigator's decision to discontinue treatment, patient withdrew consent or lost to follow-up, or study terminated by Sponsor; or until maximum of 2 years.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Expansion Cohort 3: NKTR-214 (0.010 mg/kg) + Pembro (200 mg): "NKTR-214 (0.010 mg/kg) + pembrolizumab (200 mg)
  NKTR-214: Specified dose on specified days Pembrolizumab: Specified dose on specified days"
Arm/Group | Dose Expansion Cohort 2: NKTR-214 (0.006 mg/kg) + Pembro (200 mg) | Dose Expansion Cohort 3: NKTR-214 (0.010 mg/kg) + Pembro (200 mg)
Number analyzed (Participants) | 60 | 13
Participants | 13 | 2

4. Primary Outcome: Objective Response Rate (ORR) Per Investigator's Assessment by RECIST 1.1 of NKTR-214 at a Dose of 0.006 mg/kg With Pembrolizumab and Platinum-based Chemotherapy for Dose Expansion Cohorts 4+5.
Description: ORR per Investigator's Assessment* by RECIST 1.1 for the Response Evaluable Population dose expansion Cohorts 4 +5. The Response Evaluable Population was subjects who received at least 1 dose (or partial dose) of study drug, had measurable disease (per RECIST 1.1) at baseline, and had at least 1 post-baseline assessment of tumor response.
  Objective response is the sum of confirmed complete response and confirmed partial response.
  *Efficacy endpoint for Cohort 4 +5 is per Investigator's Assessment due to the early termination of the study and incompleteness of BICR data for these cohorts.
Time Frame: Until disease progression, death, unacceptable toxicity, symptomatic deterioration, Investigator's decision to discont. treatment, patient withdrew consent or lost to follow-up, or study terminated by Sponsor; or until maximum of 2 years.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Expansion Cohorts 4/5: NKTR-214 (0.006 mg/kg) + pembrolizumab + chemotherapy
Arm/Group | Dose Expansion Cohorts 4/5
Number analyzed (Participants) | 8
Participants | 2

ADVERSE EVENTS:
Time Frame: AEs will be reported starting immediately after the patient has been administered the first dose of study drug(s) until 100 days after the last dose of all study drug(s) up to 28 months. All study treatment-related SAEs that have not resolved by the end of treatment (EOT) visit will be followed until any of the following occur (whichever comes first): the event resolves or has stabilized or event returns to baseline (if a baseline value is available), or the patient dies or is lost to follow-up.
Groups:
- Dose Expansion Cohort 3: NKTR-214 (0.010 mg/kg) + Pembro (200 mg): "NKTR-214 (0.010 mg/kg) + pembrolizumab (200 mg)
  NKTR-214: Specified dose on specified days Pembrolizumab: Specified dose on specified days
- Dose Expansion Cohorts 4/5: NKTR-214 (0.006 mg/kg) + Pembro (200 mg) + Chemotherapy: "NKTR-214 (0.006 mg/kg) + pembrolizumab (200 mg) + chemotherapy
  NKTR-214: Specified dose on specified days Pembrolizumab: Specified dose on specified days
Arm/Group | Cohort 0 (Before Protocol Amendment 5.0): NKTR-214 (0.006 mg/kg) + Pembro (200 mg) | Cohort 0 (Before Protocol Amendment 5.0): NKTR-214 (0.006 mg/kg) + Atezo (1200 mg) | Dose Optimization Cohort 1a: NKTR-214 (0.008 mg/kg) + Pembro (200 mg) | Dose Optimization Cohort 1a: NKTR-214 (0.010 mg/kg) + Pembro (200 mg) | Dose Optimization Cohort 1a: NKTR-214 (0.012 mg/kg) + Pembro (200 mg) | Dose Expansion Cohort 2: NKTR-214 (0.006 mg/kg) + Pembro (200 mg) | Dose Expansion Cohort 3: NKTR-214 (0.010 mg/kg) + Pembro (200 mg) | Dose Expansion Cohorts 4/5: NKTR-214 (0.006 mg/kg) + Pembro (200 mg) + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 4/12 | 18/23 | 3/4 | 2/7 | 5/7 | 39/75 | 5/17 | 2/17
Serious Adverse Events (participants affected / at risk) | 5/12 | 14/23 | 2/4 | 4/7 | 2/7 | 30/75 | 10/17 | 8/17
Other Adverse Events (participants affected / at risk) | 12/12 | 23/23 | 4/4 | 7/7 | 7/7 | 74/75 | 16/17 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 0 (Before Protocol Amendment 5.0): NKTR-214 (0.006 mg/kg) + Pembro (200 mg) (N=12) | Cohort 0 (Before Protocol Amendment 5.0): NKTR-214 (0.006 mg/kg) + Atezo (1200 mg) (N=23) | Dose Optimization Cohort 1a: NKTR-214 (0.008 mg/kg) + Pembro (200 mg) (N=4) | Dose Optimization Cohort 1a: NKTR-214 (0.010 mg/kg) + Pembro (200 mg) (N=7) | Dose Optimization Cohort 1a: NKTR-214 (0.012 mg/kg) + Pembro (200 mg) (N=7) | Dose Expansion Cohort 2: NKTR-214 (0.006 mg/kg) + Pembro (200 mg) (N=75) | Dose Expansion Cohort 3: NKTR-214 (0.010 mg/kg) + Pembro (200 mg) (N=17) | Dose Expansion Cohorts 4/5: NKTR-214 (0.006 mg/kg) + Pembro (200 mg) + Chemotherapy (N=17)
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 6 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bundle branch block (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Myasthenic syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 0 (Before Protocol Amendment 5.0): NKTR-214 (0.006 mg/kg) + Pembro (200 mg) (N=12) | Cohort 0 (Before Protocol Amendment 5.0): NKTR-214 (0.006 mg/kg) + Atezo (1200 mg) (N=23) | Dose Optimization Cohort 1a: NKTR-214 (0.008 mg/kg) + Pembro (200 mg) (N=4) | Dose Optimization Cohort 1a: NKTR-214 (0.010 mg/kg) + Pembro (200 mg) (N=7) | Dose Optimization Cohort 1a: NKTR-214 (0.012 mg/kg) + Pembro (200 mg) (N=7) | Dose Expansion Cohort 2: NKTR-214 (0.006 mg/kg) + Pembro (200 mg) (N=75) | Dose Expansion Cohort 3: NKTR-214 (0.010 mg/kg) + Pembro (200 mg) (N=17) | Dose Expansion Cohorts 4/5: NKTR-214 (0.006 mg/kg) + Pembro (200 mg) + Chemotherapy (N=17)
Pyrexia (General disorders) | 2 | 8 | 1 | 7 | 4 | 30 | 8 | 3
Fatigue (General disorders) | 6 | 14 | 2 | 6 | 3 | 22 | 5 | 4
Chills (General disorders) | 3 | 3 | 3 | 3 | 6 | 11 | 1 | 3
Asthenia (General disorders) | 0 | 3 | 0 | 0 | 1 | 22 | 5 | 0
Influenza like illness (General disorders) | 2 | 5 | 1 | 2 | 2 | 13 | 0 | 2
Oedema peripheral (General disorders) | 3 | 6 | 1 | 2 | 1 | 8 | 3 | 2
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0 | 1 | 5 | 1 | 0
Gait disturbance (General disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Axillary pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 8 | 2 | 7 | 3 | 18 | 6 | 10
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 1 | 4 | 2 | 16 | 5 | 7
Vomiting (Gastrointestinal disorders) | 5 | 6 | 2 | 4 | 1 | 12 | 3 | 5
Constipation (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 1 | 8 | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1 | 2 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0 | 5 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 3 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4 | 2 | 4 | 3 | 14 | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 1 | 2 | 13 | 3 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 1 | 2 | 5 | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 2 | 6 | 2 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Keratolysis exfoliativa acquired (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 2 | 2 | 2 | 2 | 1 | 12 | 4 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 2 | 3 | 12 | 2 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 2 | 2 | 10 | 2 | 2
Blood creatinine increased (Investigations) | 3 | 3 | 2 | 0 | 0 | 4 | 1 | 2
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 6 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 5 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0
Lipase increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Troponin I increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2 | 3 | 1 | 20 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 1 | 2 | 14 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 1 | 2 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 4 | 1 | 19 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0 | 0 | 8 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 1 | 0 | 5 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0 | 1 | 3 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 7 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 4 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 10 | 1 | 2 | 1 | 15 | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 2 | 9 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 0 | 5 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 2 | 5 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 2 | 0 | 1 | 2 | 3 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 0 | 2 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insulin resistance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 7 | 0 | 1 | 1 | 6 | 1 | 1
Headache (Nervous system disorders) | 3 | 3 | 1 | 2 | 1 | 5 | 3 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vasogenic cerebral oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 3 | 1 | 1 | 1 | 5 | 1 | 1
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Candida infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 0 | 1 | 13 | 2 | 2
Eosinophilia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 2 | 4 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 3 | 1 | 2 | 2 | 11 | 1 | 1
Hypertension (Vascular disorders) | 2 | 0 | 1 | 1 | 0 | 7 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 3 | 0 | 1 | 4 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 3 | 0 | 0 | 1 | 4 | 0 | 2
Depression (Psychiatric disorders) | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 2 | 1 | 1 | 0 | 9 | 4 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 2 | 1 | 1 | 0 | 10 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Androgen deficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meibomian gland dysfunction (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metamorphopsia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 0 | 3 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multiple allergies (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT03138889/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT03138889/SAP_001.pdf